CLINICAL TRIAL: NCT02273232
Title: Effects of Remote Ischemic Preconditioning on Moderate PVD Patients A Pilot Randomized Control Trial
Acronym: RIPC-PVD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, KHALID AHMED, Dr/Mr, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.A 1154
Record Dates: First submitted 2014-10-18; First posted 2014-10-23 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Arterial Diseases
Keywords: Peripheral Arterial Disease; Peripheral Vascular Disease; Claudication; Remote Ischemic Preconditioning; EQ-5D; Symptoms free distance; ABI; micro vessel formation
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Intermittent Claudication | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supervised Exercise Group (Active Comparator): All PVD patients will get the standard advice regarding exercises but this group will have a constructed exercise program under supervision of Dr. Micheál Newell who is qualified Sports and Exercise Scientist with a Doctorate degree in Integrated Biology. This include six minute walk test, Chair Stand Test and symptoms free distance.
  Interventions: Other: Supervised Exercise; Other: Standard Care
- RIPC and supervised Exercise Group (Active Comparator): This group will have structured intermitting periods of induced remote ischaemic preconditioning using standard blood pressure cuffs. The cuff will be applied for 5 minutes alternatively with 5 minutes rest to the total of 4 cycles, which needs 40 minutes per day. The RIPC group will receive an exercise program identical to the first group. The total number of days for each participant will be 28 days.
  Interventions: Other: Remote Ischemic Preconditioning; Other: Supervised Exercise; Other: Standard Care
- RIPC with Standard Care Group (Active Comparator): The patients in this group will receive standard care advice regarding exercise in addition to RIPC as in the 2nd group.
  Interventions: Other: Remote Ischemic Preconditioning; Other: Standard Care
- Control Group (Standard Care) (Sham Comparator): This group will get the standard advice regarding exercise for PVD patients and all the information available in Out patients clinic settings.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Remote Ischemic Preconditioning — Blood pressure cuff will be inflated to 200 mmhg for 5 minuets and release for 5 minuets to total of 4 cycles
  Other Names: RIPC
  Arms: RIPC and supervised Exercise Group; RIPC with Standard Care Group
Other: Supervised Exercise — constructed extra excessive for peripheral vascular diastase patients
  Arms: RIPC and supervised Exercise Group; Supervised Exercise Group
Other: Standard Care — Standard Care for peripheral vascular disease patients including advises regarding exercises

SUMMARY:
Remote ischemic Preconditioning (RIPC) is a phenomena first observed in cardio-thoracic patients in which exposing the limbs for periods of short intermittent ischemia produces protective effect on heart muscle. The concept was applied to many other parts of the body and the results are positive so far.

No human trials on this concept has been conducted in patients with peripheral vascular disease so far but applying the concept for healthy individuals shows vessels dilatation and animal trials shows degree of new vessels formation in addition to reports of symptoms improvement.

The trial candidates will be allocated blindly in 4 groups. All groups will have advice about exercise which is the standard practice now. The first group will have supervised exercise. The second group will in addition to the supervised exercise get the ischemic preconditioning with the blood pressure cuff. The third group will get the ischemic preconditioning and the fourth group will get the standard exercise advice. All candidates will have Magnetic Resonance Image Scan (MRA) for their blood vessels in the beginning of the trial and again at the end.

The effect of the RIPC (Remote ischemic Preconditioning) and exercises on patient symptoms, new vessel formation and other parameters will be recorded

DETAILED DESCRIPTION:
Peripheral vascular disease (PVD) is a major health problem, affecting approximately 20% of adults over 55 years of age and about 27 million people in North America and Europe . Most PVD is asymptomatic. Intermittent claudication is the typical clinical manifestation, developing in about 5% men aged 60 years and increases with age . For every patient with symptomatic PAD there are another three to four subjects in general population with PVD who do not meet the clinical criteria for intermittent claudication [4] . There are no precise figures for PVD's health economic impact in Ireland. In the United States, the estimated total cost of PVD exceeds $21 billion annually .

Current treatment options for non-lifestyle limiting claudication include watchful waiting, medical management, exercise training, endovascular treatment and surgical reconstruction with uncertainty regarding the optimal approach in many patients. PVD patients usually have multiple co-morbidities. Decisions regarding optimal management seek to balance the risk of intervention in patients with multiple co-morbidities, the likely benefit in terms of symptom relief and quality of life and the overall life-expectancy of these patients . There is a need for safer, non-invasive interventions which are cost-effective and acceptable to patients.

Ischemic preconditioning was first described by Murry et al, almost 30 years ago when he observed that protection was conferred on ischemic myocardium by preceding brief periods of sub lethal ischemia separated by periods of reperfusion . Subsequent experiments demonstrated that brief periods of ischemia-reperfusion in any tissue conferred protection on any other tissue exposed to a significant ischemic insult. For example, brief periods of skeletal muscle ischemia-reperfusion confers protection on the heart. This phenomenon is referred to as remote ischemic preconditioning (RIPC)

Clinical trials in cardiac surgery and percutaneous coronary intervention suggest that RIPC reduces cardiac injury, critical care stay and inotropes use. However, the effects of preconditioning in peripheral vascular disease patients remain largely un evaluated, apart from some small studies on symptomatic relief and the exercise induced preconditioning effect . Remote preconditioning affects blood supply in other limbs. Enko et al demonstrated that intermittent arm ischemia by applying 3 cycles of 200mmHg pressure for 5 minutes, followed by 5 minutes of reperfusion produced dilatation of the contralateral brachial artery in healthy individuals. In a more recent study, Karakyoun et al evaluated RIPC and direct preconditioning in a rat model of critical limb ischemia. Iliac artery ligation was used to create critical limb ischemia in the rats. Both direct preconditioning (intermittent tourniquet application in the ischemic limb) and RIPC (intermittent tourniquet application on the contralateral leg) produced significant increases in perfusion and microvasculature density in the ischemic limb with true new blood vessels formation in both direct the IC and RIPC groups .

The investigators hypothesize that remote preconditioning as an adjunct to exercise therapy or alone could stimulate greater microvessel formation in the legs of claudication patients, improving clinical outcomes in terms of symptoms and delayed complications. It may provide a new non-invasive option for PVD patients.

Sampling Frame All peripheral vascular disease patients referred to UCHG (University Collage Hospital Galway) OPD (Out Patients) in addition to inpatients during trial period will be actively searched to identify medical profiles which fulfill the trial criteria. Recruitment for the trial will be stopped at 15 months of 24 months' time frame.

Trial Design Patients referred to vascular service OPDs (out patients) with claudication symptoms for the first time are usually assessed a by consultant or specialty registrar. Further investigations and course of management depends mainly on their symptoms and co morbidities. Many end up with diagnosis of peripheral vascular disease. From this group in addition to in patients group those with moderate peripheral vascular disease i.e., Rutherford stage 2 and Fontaine stage 2a. Will be recruited

The target number will be 40 patients divided into 4 groups. All groups candidate will undergo base line assessment which include history, examination, MRA and ABIs. The candidates will be randomized into:

Supervised Exercise Group:

All PVD patients will get the standard advice regarding exercises but this group will have a constructed exercise program under supervision of Dr. Micheál Newell who is qualified Sports and Exercise Scientist with a Doctorate degree in Integrated Biology. This include six minute walk test, Chair Stand Test and symptoms free distance.

RIPC and supervised Exercise Group:

This group will have structured intermittent periods of induced remote ischemic preconditioning using standard blood pressure cuffs. The cuff will be applied for 5 minutes alternatively with 5 minutes rest to the total of 4 cycles, which needs 40 minutes per day. The RIPC group will receive an exercise program identical to the first group. The total number of days for each participant will be 30 days.

RIPC with Standard Care Group:

The patients in this group will receive standard care advice regarding exercise in addition to RIPC as in the 2nd group.

Control Group (Standard Care):

This group will get the standard advice regarding exercise for PVD patients and all the information available in OPD settings.

Sample Size:

The trial will be a pilot study to obtain preliminary data and evaluate the need for full-scale trial hence there is no human trial in this particular area so far. The initial target will be 40 patients distributed in 4 groups of 10 patient each.

Randomization Age and DM (Diabetes Mellitus ) are associated with many comorbidities. Randomization will be stratified for these two confounders.

All trial candidates will have unique numbers to identify them and conceal their identity. Patients files will be locked in trial office with one person access and each candidate will get their numbers in sequential way according to their allocation.

Projected recruitment Galway University hospital provides vascular services for a population of approximately 750000 served by the West-North West Hospitals Group. The patients for the trial will be actively recruited from out patients clinics, in patients and GP clinics by sending letters to GPs ( General practitioners ) about the trial. Information about the trial will be given to all vascular team including criteria for selection and exclusion. Those who qualified will be counselled by the trial team and consented if the agree to join. The target of 40 patients should be achievable within the recruitment window.

Patient recruitment & consent Eligible candidates will be given all the information about the trial in written and verbal explanation for all the steps. Patients who are willing to take part will be asked to provide written informed consent. Three copies of the consent form will be signed: one for the patient, one for the patient's clinical notes file and a one copy for the patient's trial folder.

Data collection Demographic and clinical data of eligible candidates who agree to participate will be collected. The candidates will be assign a trial number identifier after informed consent is signed and no personal information will be available on the data entry sheets. The original data-entry proforma will be retained together with a copy of the consent form in the trial office with other trial documents in the trial office in CSI( Clinical Science Institute) building. The code key for the trial numbers will be limited to the Chief Investigator. Encrypted back up copy will be prepared at the end of each data entry and will be kept looked separately. All data will be retained in the care of the principal investigator for a period of five years from the closure of the trial.

Statistical analysis The statistical analysis with respect to the primary and secondary outcomes will be performed by a trial team member blinded to trial allocation. The cost-effectiveness analysis will be performed under the supervision of the trial health-economist (to be confirmed). This is a pilot study the results will identify if there is a need for larger trial.

Trial monitoring Day-to-day management of the trial will be the responsibility of the trial manager, supervised by the principal investigator. A meeting will be held every two weeks between the trial manager and the principal investigator to monitor recruitment, data collection etc.

ELIGIBILITY:
Inclusion Criteria:

1. Known moderate PVD
2. New claudication patient with Rutherford stage 2 and Fontaine stage 2a symptoms

Exclusion Criteria:

1. Known upper limb PVD
2. Severe cardiac condition
3. Risk classification for exercise training: class C and above
4. Severe respiratory condition
5. Previous history of upper limb deep vein thrombosis
6. Patients on glibenclamide or nicorandil- May affect RIPC
7. Raynaud's Disease
8. Contra indications for MRA
9. Pregnancy
10. Previous major limb amputation affect ability to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Symptoms free distance | 30 days
  Distance which patient can walk without pain at the beginning and the end of the trial will be compared and compared cross groups
ABI -Ankle-Brachial Index Test | 30 days
  ABI measured at the beginning and the end of the trial comparing pre and post results in all groups will be analysed
6-minute walk test | 30 days
  The standard Test (american college of rheumatology) results will be measured pre and post trial to evaluate any change in functional exercise capacity
EQ-5D quality of life measures | 6 months
  EQ-5D questionnaire will be used as slandered Quality of life assessment tool post trial for candidates a cross groups - http://www.euroqol.org/

SECONDARY OUTCOMES:
Effects on BP (Blood Pressure ) | 30 days
  changes in BP before after intervention will be evaluated
% changes in ABI | 30 days
  Ankle-Brachial Index percentage changes will be calculated comparing ABI measurement before and after Trial
Minor amputations | 30 days
  Minor amputations (digits) due to disease will be detailed in percentage among groups
Progress for amputation during trial | 30 days
  Record of Progress for amputation during trial - Amputations in the previous outcome will be excluded
Progression of Rutherford classification | 30 days
  record of claudication distance Progression during trial using Rutherford classification

CONTACTS AND LOCATIONS:
Overall Officials: Stewart E Walsh, Professor, Principal Investigator — NUIG
Locations (1):
- University Collage Hospital Galway, Galway, Co Galway, Ireland

REFERENCES:
- [Result] Andreozzi GM, Leone A, Laudani R, Deinite G, Martini R. Acute impairment of the endothelial function by maximal treadmill exercise in patients with intermittent claudication, and its improvement after supervised physical training. Int Angiol. 2007 Mar;26(1):12-7. PMID 17353883
- [Result] Birnbaum Y, Hale SL, Kloner RA. Ischemic preconditioning at a distance: reduction of myocardial infarct size by partial reduction of blood supply combined with rapid stimulation of the gastrocnemius muscle in the rabbit. Circulation. 1997 Sep 2;96(5):1641-6. doi: 10.1161/01.cir.96.5.1641. PMID 9315559
- [Result] Capecchi PL, Pasini FL, Cati G, Colafati M, Acciavatti A, Ceccatelli L, Petri S, de Lalla A, Di Perri T. Experimental model of short-time exercise-induced preconditioning in POAD patients. Angiology. 1997 Jun;48(6):469-80. doi: 10.1177/000331979704800601. PMID 9194532
- [Result] Dickson EW, Porcaro WA, Fenton RA, Heard SO, Reindhardt CP, Renzi FP, Przyklenk K. "Preconditioning at a distance" in the isolated rabbit heart. Acad Emerg Med. 2000 Apr;7(4):311-7. doi: 10.1111/j.1553-2712.2000.tb02228.x. PMID 10805617
- [Result] Dormandy J, Heeck L, Vig S. Intermittent claudication: a condition with underrated risks. Semin Vasc Surg. 1999 Jun;12(2):96-108. PMID 10777236
- [Result] Enko K, Nakamura K, Yunoki K, Miyoshi T, Akagi S, Yoshida M, Toh N, Sangawa M, Nishii N, Nagase S, Kohno K, Morita H, Kusano KF, Ito H. Intermittent arm ischemia induces vasodilatation of the contralateral upper limb. J Physiol Sci. 2011 Nov;61(6):507-13. doi: 10.1007/s12576-011-0172-9. Epub 2011 Sep 8. PMID 21901641
- [Result] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Result] Fowkes FG, Housley E, Cawood EH, Macintyre CC, Ruckley CV, Prescott RJ. Edinburgh Artery Study: prevalence of asymptomatic and symptomatic peripheral arterial disease in the general population. Int J Epidemiol. 1991 Jun;20(2):384-92. doi: 10.1093/ije/20.2.384. PMID 1917239
- [Result] Hankey GJ, Norman PE, Eikelboom JW. Medical treatment of peripheral arterial disease. JAMA. 2006 Feb 1;295(5):547-53. doi: 10.1001/jama.295.5.547. PMID 16449620
- [Result] Karakoyun R, Koksoy C, Yilmaz TU, Altun H, Banli O, Albayrak A, Alper M, Sener Z. The angiogenic effects of ischemic conditioning in experimental critical limb ischemia. Eur J Vasc Endovasc Surg. 2014 Feb;47(2):172-9. doi: 10.1016/j.ejvs.2013.11.001. Epub 2013 Nov 11. PMID 24333045
- [Result] Layden J, Michaels J, Bermingham S, Higgins B; Guideline Development Group. Diagnosis and management of lower limb peripheral arterial disease: summary of NICE guidance. BMJ. 2012 Aug 8;345:e4947. doi: 10.1136/bmj.e4947. No abstract available. PMID 22875949
- [Result] Mahoney EM, Wang K, Keo HH, Duval S, Smolderen KG, Cohen DJ, Steg G, Bhatt DL, Hirsch AT; Reduction of Atherothrombosis for Continued Health (REACH) Registry Investigators. Vascular hospitalization rates and costs in patients with peripheral artery disease in the United States. Circ Cardiovasc Qual Outcomes. 2010 Nov;3(6):642-51. doi: 10.1161/CIRCOUTCOMES.109.930735. Epub 2010 Oct 12. PMID 20940249
- [Result] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Result] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Result] Walsh SR, Tang TY, Kullar P, Jenkins DP, Dutka DP, Gaunt ME. Ischaemic preconditioning during cardiac surgery: systematic review and meta-analysis of perioperative outcomes in randomised clinical trials. Eur J Cardiothorac Surg. 2008 Nov;34(5):985-94. doi: 10.1016/j.ejcts.2008.07.062. Epub 2008 Sep 9. PMID 18783958